CLINICAL TRIAL: NCT03870737
Title: Four-week Open-trial Extension Study of Trigeminal Nerve Stimulation (TNS) for Youth Previously Randomized to Sham in a Double-Blind Trial
Brief Title: Four-week Open-trial Extension TNS for ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James McGough, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIH R34MH101282; R34MH101282 (NIH)
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Results first posted 2019-04-26 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; neuromodulation; trigeminal nerve stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active TNS (Experimental): Participants who previously underwent screening and determination of eligibility in a double-blind sham-controlled trial of TNS for ADHD, and randomized to sham, will be offered upon unblinding at the end of the 5-week controlled trial to receive 4-weeks open treatment with the active TNS condition.
  Interventions: Device: Active TNS

INTERVENTIONS:
Device: Active TNS — Participants will receive 4-weeks nightly treatment with active TNS. Positive responders will be invited to participate in 12-month open-extension study.
  Other Names: Trigeminal Nerve Stimulation; Monarch eTNS SystemTM (NeuroSigma, Inc., Los Angeles CA

SUMMARY:
The purpose of this study will be to offer children previously randomized to sham treatment in a 5-week double-blind sham controlled study of Trigeminal Nerve Stimulation for ADHD (NCT02155608) an opportunity to receive 4-weeks active TNS treatment.

DETAILED DESCRIPTION:
This study will enroll participants with ADHD who previously participated in a 5-week sham-controlled investigation of Trigeminal Nerve Stimulation as a treatment for ADHD, and who were randomized to the sham condition.

In the double-blind trial (NCT02155608), children ages 8-12 years undergo study screening and if eligible begin 4 weeks nightly treatment with active or sham TNS administered nightly during sleep. At the conclusion of the 4-week trial, all interventions (both active and sham TNS) are discontinued with blinding remaining in place for an additional week to assess possible residual treatment effects. Participants' randomized condition is unblinded at Week 5.

All participants randomized to sham in the double-blind trial are invited to participate in a 4-week open-trial of TNS to allow all participants the opportunity to benefit from the active intervention.

During this 4-week open-extension trial, interested participants will receive nightly active TNS during sleep. The final study visit (Visit 5) of the double-blind study will serve as baseline for this open-extension. Participants will return for clinic assessments at Weeks 2 and 4. Participants who achieve clinically significant improvement from active TNS over the 4-week open trial will be invited to receive a year of nightly active-TNS therapy as part of a 12-month extension study.

ELIGIBILITY:
Inclusion Criteria:

* male and female children ages 8-12 with DSM-5 ADHD, and current presentation, as determined by KSADS and clinical interview
* participated in a previous randomized, double-blind, sham-controlled trial of TNS for ADHD, and randomized to the sham condition.
* parents able and willing to monitor proper use of the TNS device and complete all required rating scales
* parent and participants able to compete study rating scales and other measures in English

Exclusion Criteria:

* currently requiring any medication with CNS effects

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J. McGough, M.D., Principal Investigator — University of California, Los Angeles; Sandra K. Loo, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active TNS
Started | 22
Completed | 20
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Active TNS
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.39 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
ADHD-Rating Scale Total Score [Mean (Standard Deviation); unit: score a scale] — A dimensional rating of ADHD symptoms, with scores ranging from 0 to 54, with higher scores signifying worse severity.
  score a scale | 20.91 (8.76)
Clinical Global Impression - Severity [Count of Participants; unit: Participants] — A categorical measure of severity ranging from 1 ("Normal, not at all ill") to 7 (Among the most seriously ill).
  Participants
    3 (Mildly ill) | 2
    4 (Moderately ill) | 4
    5 (Markedly ill) | 16

OUTCOME MEASURES:

1. Primary Outcome: ADHD-IV Rating Scale (ADHD-RS)
Description: A dimensional rating of ADHD symptoms, with scores ranging from 0 to 54, with higher scores signifying worse severity.
Time Frame: Change over Baseline, Week 2, Week 4.
Population: Some participants lost to follow up.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active TNS
Number analyzed (Participants) | 22
score on a scale
  Baseline | 28.50 (1.74)
  Week 2 | 20.91 (1.74)
  Week 4: number analyzed (Participants) | 20
  Week 4 | 18.63 (1.85)
Statistical Analysis 1: Comparison: Active TNS; Outcomes fitted via a mixed effects model with time as predictor; Test type: Superiority; p < .0001, Mixed Models Analysis; Time: F = 24.81, df = 1/40

2. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: Categorical measure indicating degree improved or not improved compared with global functioning at baseline in the preceding double-blind trial. The base CGI-I scale is a 7-point measure that requires the investigator to assess how much the condition has improved or worsened compared to baseline prior to initiation of treatment. Ratings are (1) very much improved; (2) much improved; (3) minimally improved; (4) no change; (5) minimally worse; (6) much worse; (7) very much worse. For purposes of analysis, the measure is dichotomized such that scores <= 2 signify "improved" and scores > 2 signify "not improved."
Time Frame: Change over Baseline, Week 2, Week 4
Population: Some participants lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Active TNS
Number analyzed (Participants) | 22
Participants
  Week 2: Improved | 11
  Week 2: Not Improved | 11
  Week 4: number analyzed (Participants) | 20
  Week 4: Improved | 12
  Week 4: Not Improved | 8

3. Secondary Outcome: Height
Description: A dimensional measure assessed in cm.
Time Frame: Change over Baseline, Week 2, Week 4
Population: Some participants lost to follow up.
Measure: Least Squares Mean (Standard Error); unit: cm.
Arm/Group | Active TNS
Number analyzed (Participants) | 22
cm.
  Baseline | 140.19 (2.02)
  Week 2 | 140.49 (2.02)
  Week 4: number analyzed (Participants) | 20
  Week 4 | 140.92 (2.02)
Statistical Analysis 1: Comparison: Active TNS; Outcome was fitted using a mixed model with time as predictor; Test type: Superiority; p = .02, Mixed Models Analysis; Time: F = 5.78, df = 1/39

4. Secondary Outcome: Weight
Description: A dimensional measure assessed in kg.
Time Frame: Change over Baseline, Week 2, Week 4
Population: Some participants lost to follow up.
Measure: Least Squares Mean (Standard Error); unit: kg.
Arm/Group | Active TNS
Number analyzed (Participants) | 22
kg.
  Baseline | 34.19 (1.53)
  Week 2 | 34.61 (1.53)
  Week 3: number analyzed (Participants) | 20
  Week 3 | 34.91 (1.53)
Statistical Analysis 1: Comparison: Active TNS; Outcome was fitted using a mixed model with time as predictor; Test type: Superiority; p = .0005, Mixed Models Analysis; Time: F = 14.28, df = 1/39

5. Secondary Outcome: Systolic Blood Pressure
Description: A dimensional measure assessed in mm HG.
Time Frame: Change over Baseline, Week 2, Week 4
Population: Some participants lost to follow up.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Active TNS
Number analyzed (Participants) | 22
mm Hg.
  Baseline | 107.27 (2.22)
  Week 2 | 109.83 (2.30)
  Week 4: number analyzed (Participants) | 20
  Week 4 | 107.78 (2.30)
Statistical Analysis 1: Comparison: Active TNS; Outcome was fitted using a mixed model with time as predictor; Test type: Superiority; p = .67, Mixed Models Analysis; Time: F = .19, df = 1/39

6. Secondary Outcome: Diastolic Blood Pressure
Description: A dimensional measure assessed in mm HG.
Time Frame: Change over Baseline, Week 2, Week 4
Population: Some participants lost to follow up.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Active TNS
Number analyzed (Participants) | 22
mm Hg.
  Baseline | 59.41 (1.91)
  Week 2 | 58.36 (1.99)
  Week 4: number analyzed (Participants) | 20
  Week 4 | 60.51 (1.99)
Statistical Analysis 1: Comparison: Active TNS; Outcome was fitted using a mixed model with time as predictor; Test type: Superiority; p = .76, Mixed Models Analysis; Time: F = .08, df = 1/39

7. Secondary Outcome: Pulse
Description: A dimensional measure assessed in heart beats per minute.
Time Frame: Change over Baseline, Week 2, Week 4
Population: Some participants lost to follow up.
Measure: Least Squares Mean (Standard Error); unit: heart beats per minute.
Arm/Group | Active TNS
Number analyzed (Participants) | 22
heart beats per minute.
  Baseline | 75.81 (2.76)
  Week 2 | 77.04 (2.81)
  Week 4: number analyzed (Participants) | 20
  Week 4 | 76.11 (2.81)
Statistical Analysis 1: Comparison: Active TNS; Outcome was fitted using a mixed model with time as predictor; Test type: Superiority; p = .80, Mixed Models Analysis; Time: F = .06, df = 1/39

8. Other Pre Specified Outcome: Conners Global Index - Parent Report
Description: Parent completed dimensional rating of ADHD symptoms,with score range from 0- 30, and higher scores indicating more severe symptoms.
Time Frame: Change over Baseline and weekly for 4-week trial
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Conners Global Index - Teacher Report
Description: Teacher completed dimensional rating of ADHD symptoms,with scores ranging from 0-30, and higher scores indicating more severe symptoms.
Time Frame: Change over Baseline and weekly for 4-week trial
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Affective Reactivity Index (ARI-C) Child
Description: A child-completed dimensional measure of emotional reactivity,with scores ranging from 0-12, and higher scores indicating greater severity.
Time Frame: Change over Baseline, Week 4
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Affective Reactivity Index (ARI-P) Parent
Description: A parent-completed dimensional measure of emotional reactivity, with scores ranging from 0-12, and higher scores indicating greater severity.
Time Frame: Change over Baseline, Week 4
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Children's Sleep Habits Questionnaire (CSHQ)
Description: A parent-completed 33-item scale to assess sleep related problems. Total scores range from 33 to 99 divided among 8 sub scales , with higher scores indicating more severe difficulties.
Time Frame: Change over Baseline and weekly for 4-week trial
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Multidimensional Anxiety Scale for Children (MASC) - Child Report
Description: A child-completed rating of child anxiety, with scores ranging from 0-300, and higher scores indicating greater severity.
Time Frame: Change over Baseline and Week 4
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Multidimensional Anxiety Scale for Children (MASC) - Parent Report
Description: A parent-completed rating of child anxiety, with scores ranging from 0-300, and higher scores indicating greater severity.
Time Frame: Change over Baseline and Week 4
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Children's Depression Rating Scale - Revised (CDRS-R)
Description: A clinician-completed dimensional measure of childhood mood symptoms obtained from parent and child interview, with range of scores from 17 to 113, and higher scores indicating more severe depression. A score >= 40 suggests depression; scores <= 28 defines remission.
Time Frame: Change over Baseline and Week 4
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Behavior Rating Inventor of Executive Functioning (BRIEF)
Description: A parent completed rating of child executive function. Comprises 5 sub scales that measure various measures of behavior and cognition. Raw scores on each measure are converted to T scores ranging from 28 to 103, with higher scores indicating greater difficulties.
Time Frame: Change over Baseline and weekly during 4-week trial
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: standard instrument to assess potential suicidality with dichotomous scores (0 = absent; 1 = present) to rate various components of suicidal ideation and behavior. Data derived are summarized under Adverse Event Reporting.
Time Frame: Baseline and weekly during 4-week trial
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data were collected over the 4-week open trial, beginning at baseline and then at weeks 2 and 4.
Description: Adverse events were solicited via a structured side effects questionnaire and open inquiry completed at each assessment point
Arm/Group | Active TNS
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 14/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TNS (N=22)
Stomachache (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (5)
Trouble hearing (Ear and labyrinth disorders) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Headache (Nervous system disorders) | 1 (1)
Drowsy (General disorders) | 2 (3)
Fatigue (General disorders) | 1 (1)
Trouble sleeping (Psychiatric disorders) | 2 (3)
Nightmares (Psychiatric disorders) | 1 (1)
Hyperactive (Psychiatric disorders) | 8 (13)
Feels strange (Psychiatric disorders) | 1 (1)
Difficulty finding words (Nervous system disorders) | 1 (1)
Apathy (Psychiatric disorders) | 2 (2)
Suicidal ideation with active plan and intent (Psychiatric disorders) | 0 (0) — Based on the Columbia Suicide Severity Rating Scale (C-SSRS)
Suicidal ideation with some intent (Psychiatric disorders) | 0 (0) — Based on the Columbia Suicide Severity Rating Scale (C-SSRS)
Active suicidal ideation without intent (Psychiatric disorders) | 0 (0) — Based on the Columbia Suicide Severity Rating Scale (C-SSRS)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2015-04-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03870737/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03870737/Prot_SAP_002.pdf